CLINICAL TRIAL: NCT05137912
Title: Neoadjuvant Immunotherapy in Advanced NSCLC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: e4c2e8edac362acab7123654b9e734
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer, Non-small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Immunotherapy — Patients within this intervention group will be histologically confirmed to have resectable non small cell lung cancer with stage II-IIIA.
  Patients may receive single agent immunotherapy or immunotherapy combined with chemotherapy.

SUMMARY:
A number of clinical trials have demonstrated the efficacy of immunotherapy prior as neoadjuvant therapy. This study evaluates whether said neoadjuvant immunotherapy may improve improve progression free survival in NSCLC. One such example would be to evaluate either single agent or an immunotherapy combination with chemotherapy. Following this, analysis of biomarkers will be conducted to provide personalization in one's regimen.

DETAILED DESCRIPTION:
A number of clinical trials have demonstrated the efficacy of immunotherapy prior as neoadjuvant therapy. This study evaluates whether said neoadjuvant immunotherapy may improve improve progression free survival in NSCLC. [The Power Life Sciences Investigative Team](https://www.withpower.com) is running a study to evaluate either single agent or an immunotherapy combination with chemotherapy. Patients can contact a site administrator via the information below, or enroll directly via <a href="https://www.withpower.com/trial/phase-4-2019-e67c1">https://www.withpower.com/trial/phase-4-2019-e67c1</a>. Following this, analysis of biomarkers will be conducted to provide personalization in one's regimen.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 Years of Age
* Informed consent is provided
* Histologically confirmed resectable non-small cell lung cancer with stage II-IIIA (TNM 8th edition)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Epidermal growth factor receptor (EGFR) mutation negative and anaplastic lymphoma kinase (ALK) translocation negative

Exclusion Criteria:

* EGFR mutation positive and ALK translocation positive
* Active central nervous system (CNS) metastases
* Autoimmune diseases
* Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Patients with interstitial lung disease will not be included if they have symptomatic interstitial lung disease (ILD) - Grade 3-4
* Women who are breast feeding or pregnant
* Sexually active women or men of childbearing potential who are not willing to use an effective contraceptive method during the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stage IIA-IIIA NSCLC
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response | 12 Weeks
  To evaluate the major pathological response (MPR) rate of participants

SECONDARY OUTCOMES:
Objective Response Rate | 12 Weeks
  Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST)
MPR based on diverse PD-L1 expression | 12 Weeks
  Percentage of Participants with Major Pathologic Response Rates For Programmed Death Ligand 1 (PD-L1)-Positive Versus PD-L1-Negative Participants
Progression Free Survival | 12 Weeks
  Progression Free Survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — [Power Life Sciences Inc.](www.withpower.com)
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jiang L, Huang J, Jiang S, Rong W, Shen Y, Li C, Tian Y, Ning J, Chen X, Yang Y, Ding Z, Li Z, Luo Q. The surgical perspective in neoadjuvant immunotherapy for resectable non-small cell lung cancer. Cancer Immunol Immunother. 2021 Aug;70(8):2313-2321. doi: 10.1007/s00262-021-02847-1. Epub 2021 Jan 29. PMID 33512555
- [Background] Broderick SR. Adjuvant and Neoadjuvant Immunotherapy in Non-small Cell Lung Cancer. Thorac Surg Clin. 2020 May;30(2):215-220. doi: 10.1016/j.thorsurg.2020.01.001. PMID 32327180
- [Background] Gutierrez-Sainz L, Cruz-Castellanos P, Higuera O, de Castro-Carpeno J. Neoadjuvant Chemoimmunotherapy in Patients with Resectable Non-small Cell Lung Cancer. Curr Treat Options Oncol. 2021 Aug 23;22(10):91. doi: 10.1007/s11864-021-00885-6. PMID 34424417
- See also: Participating Patient Terms of Service — https://www.withpower.com/terms-of-service
- See also: Immunotherapy As Neoadjuvant Therapy For Non Small Cell Lung Cancer — https://www.withpower.com/trial/phase-4-2019-e67c1
- See also: Patient Support Line — https://www.withpower.com/contact-us

DOCUMENTS (1):
  • Informed Consent Form (2021-11-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT05137912/ICF_000.pdf